CLINICAL TRIAL: NCT05990504
Title: The Effect of Dural Puncture Epidural Block Technique on the Effectiveness and Safety of Labor Analgesia
Acronym: DPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zongxun Lin (Other)
Responsible Party: Sponsor-Investigator, Zongxun Lin, Principal Investigator, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dural Puncture Epidural
Record Dates: First submitted 2023-04-21; First posted 2023-08-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Labor Analgesia
Keywords: labor analgesia; delivery woman; neonate; Effectiveness; Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dural Puncture Epidural Group (Experimental): Dural Puncture Epidural is a new type of labor analgesia technology.
  Interventions: Device: ultrasound real-time guidance combined with Dural Puncture Epidural Labor Anagesia
- Epidural Group (Active Comparator): Epidural is a traditional labor analgesia technique.
  Interventions: Device: ultrasound real-time guidance combined with Epidural Labor Anagesia

INTERVENTIONS:
Device: ultrasound real-time guidance combined with Dural Puncture Epidural Labor Anagesia — Dural Puncture Epidural is a clinical improvement of Combined Spinal-Epidural and is widely used in Maternal. The implementation step is to complete the epidural puncture, temporarily do not place a tube, puncture the dura mater with a subarachnoid anesthesia needle, but do not directly inject drugs into the subarachnoid space, and then leave an epidural catheter for administration according to epidural block.
  Arms: Dural Puncture Epidural Group
Device: ultrasound real-time guidance combined with Epidural Labor Anagesia — Epidural is a traditional labor analgesia technique.
  Arms: Epidural Group

SUMMARY:
Dural Puncture Epidural is a clinical improvement of Combined Spinal-Epidural and is widely used in Maternal.Dural Puncture Epidural Technique improves Labor Analgesia Quality And Safety By Increasing Drug Permeation.This study combines ultrasound real-time guidance technology. This technology ensures the accuracy of intervertebral space positioning and puncture success rate through operational visualization, and reduces the impact of operator proficiency on research results.

DETAILED DESCRIPTION:
Dural Puncture Epidural is a clinical improvement of Combined Spinal-Epidural and is widely used in Maternal. The implementation step is to complete the epidural puncture, temporarily do not place a tube, puncture the dura mater with a subarachnoid anesthesia needle, but do not directly inject drugs into the subarachnoid space, and then leave an epidural catheter for administration according to epidural block. The theoretical basis is that anesthetic drugs can originally penetrate into the subarachnoid space from the epidural space through a complete spinal dura, and the puncture hole formed by spinal dura puncture facilitates this process.After injecting high volume anesthetic drugs into the epidural space, the pressure increases, and the drug penetrates from the epidural space through the puncture hole along a pressure gradient to the subarachnoid space, thereby enhancing the effect of labor analgesia.Dural Puncture Epidural also has the advantage of verifying that the epidural needle is in the middle of the epidural space again, thereby reducing the incidence of epidural catheter insertion failure or deviation to one side.This study combines ultrasound real-time guidance technology. This technology ensures the accuracy of intervertebral space positioning and puncture success rate through operational visualization, and reduces the impact of operator proficiency on research results.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) Class I or II;
2. Single healthy pregnancy;
3. Head showing first;
4. 37 to 41 weeks;
5. The labor process is active, and the cervix dilates<5cm;
6. Require epidural labor analgesia;
7. Volunteer to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Presence of pregnancy diseases, such as pregnancy hypertension, pre eclampsia, pregnancy diabetes;
2. Contraindications to intraspinal analgesia: 1) Central nervous system diseases. 2) Infection or septicemia at the puncture site. 3) Coagulation dysfunction;
3. Known cases of fetal malformation or increased risk of cesarean section, such as a history of uterine rupture;
4. Persons with a history of mental illness, hysteria, epilepsy, etc. who cannot cooperate.
5. Patients with long-term use of opioids, steroids, and chronic pain.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
The incidence of NICHD category elevation from baseline | From the baseline assessment (pre-analgesia) through delivery(assessed up to 24 hours).
  NICHD (National Institute of Child Health and Human Development) Fetal Heart Tracing Classification: Category I (normal), Category II (indeterminate), Category III (abnormal). A higher category (e.g., III vs. I) indicates a less reassuring fetal status.

SECONDARY OUTCOMES:
Distribution of NICHD categories (I, II, III) | From the baseline assessment (pre-analgesia) through delivery(assessed up to 24 hours).
  NICHD (National Institute of Child Health and Human Development) Fetal Heart Tracing Classification: Category I (normal), Category II (indeterminate), Category III (abnormal). A higher category (e.g., III vs. I) indicates a less reassuring fetal status.
Fetal heart rate | From the baseline assessment (pre-analgesia) through delivery(assessed up to 24 hours).
  Assess fetal heart rate(time-weighted mean derived from area under the curve calculation).
Duration of individual uterine contractions | From the baseline assessment (pre-analgesia) through delivery(assessed up to 24 hours).
  Time-weighted mean duration of individual uterine contractions, derived from area under the curve (AUC) calculation
Incidence of hypertonus | From the baseline assessment (pre-analgesia) through delivery(assessed up to 24 hours).
  defined as a single contraction lasting >2 minutes
Incidence of tachysystole | From the baseline assessment (pre-analgesia) through delivery(assessed up to 24 hours).
  defined as >5 contractions per 10 minutes
Uterine contraction frequency | From the baseline assessment (pre-analgesia) through delivery(assessed up to 24 hours).
  Time-weighted mean uterine contraction frequency, derived from area under the curve (AUC) calculation
Incidence of asymmetric block | During the labor analgesia period (assessed up to 24 hours)
  defined as a ≥2-dermatome difference between left and right sides
Sensory blockade level | During the labor analgesia period (assessed up to 24 hours)
  Sensory blockade level was assessed by loss of cold sensation using an alcohol swab. The sensory level was determined and recorded in accordance with anatomical landmarks: pubic symphysis (T12), umbilical region (T10), hypochondrium (T8), xiphoid process (T6), nipple line (T4), and subclavian region (T2).
Time to analgesia onset | Within 30 minutes after initial drug administration
  The time from initial drug administration to the first documented pain Visual Analogue Scale (VAS) score ≤ 30 mm. Visual Analogue Scale（scale title=Visual Analogue Scale，Total score=0-10,0=no pain,10=worst possible pain）
Number of patient-controlled analgesia (PCA) demands | Through the completion of labor analgesia (assessed from initiation to delivery, up to 24 hours).
  Number of patient-controlled analgesia (PCA) demands(Press the PCA button when the patient feels pain)
Motor blockade assessed by the Modified Bromage Score | During the labor analgesia period (assessed up to 24 hours)
  Modified Bromage Score: 0 = full flexion of knees and ankles, 1 = partial flexion of knees, full flexion of ankles, 2 = inability to flex knees and partial flexion of ankles, and 3 = inability to flex knees and ankles.
Sensory blockade at the second sacral dermatome (S2) | During the labor analgesia period (assessed up to 24 hours)
  Sensory blockade at the second sacral dermatome (S2) (bilateral, unilateral, none)
Visual Analogue Scale | Through the completion of labor analgesia (assessed from initiation to delivery, up to 24 hours).
  Time-weighted mean pain Visual Analogue Scale (VAS) score, derived from area under the curve (AUC) calculation; Visual Analogue Scale（scale title=Visual Analogue Scale，Total score=0-10,0=no pain,10=worst possible pain）
Procedure-related complications of labor analgesia | From the time of the analgesia procedure until the completion of the study-specific follow-up period(assessed up to 1 week)
  Accidental dural puncture with an epidural needle
Cesarean delivery rate | At delivery
  Cesarean delivery rate among parturients receiving labor analgesia
Neonatal Apgar scores | At 1, 5, and 10 minutes after birth
  The Apgar score is a standardized assessment of newborn viability, ranging from 0 to 10. Scores are typically interpreted as: 0-3 indicating a need for urgent resuscitation, 4-6 indicating a need for some resuscitative measures, and 7-10 generally considered reassuring. In this study, Apgar scores are assessed at 1, 5, and 10 minutes after birth.
Fetal heart rate variability | Baseline period (prior to analgesia initiation) and the analgesia period (from initiation to fetal delivery)(assessed up to 24 hours).
  Assess fetal heart: Fetal heart rate variability (absent, minimal, moderate, marked)
Fetal Heart Rate decelerations | Baseline period (prior to analgesia initiation) and the analgesia period (from initiation to fetal delivery)(assessed up to 24 hours).
  Assess fetal heart: Fetal heart rate decelerations (early, late, variable)
Clinician interventions | The analgesia period (from initiation to fetal delivery)(assessed up to 24 hours).
  Clinician interventions (Analgesic Regimen Adjustments, Epidural Catheter Manipulations, Re-puncture)
Local anesthetic consumption | The analgesia period (from initiation to fetal delivery)(assessed up to 24 hours).
  Per-minute local anesthetic consumption and Total local anesthetic consumption
The duration of each stage of labor | From labor onset to delivery of placenta(assessed up to 24 hours).
  The duration of the first, second, third, and total stages of labor
Maternal body temperature | Pre-analgesia and at delivery
  Maternal body temperature (pre-analgesia and at delivery)
Side effects and complications of labor analgesia | From analgesia initiation until 72 hours after delivery (assessed up to 72 hours)
  Incidence of lower limb numbness, Incidence of urinary retention, Incidence of nausea and vomiting, Incidence of postpartum headache
Indications for cesarean delivery | At the time of cesarean delivery
  Indications for cesarean delivery (non-reassuring fetal heart rate, arrest of descent, maternal indications, other)
Anesthetic technique for cesarean delivery | At the time of cesarean delivery
  Anesthetic technique for cesarean delivery (epidural top-up, re-puncture combined spinal-epidural, general anesthesia)(Exploratory analysis added post-hoc based on reviewer feedback during the peer-review process for manuscript [Anesthesiology Research and Practice, Manuscript ID: 1197441])

CONTACTS AND LOCATIONS:
Overall Officials: Zongxun Lin, Master, Principal Investigator — Fujian Provincial Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No